CLINICAL TRIAL: NCT05141981
Title: Sarcopenia and Its Associated Factors Among Hip Fracture Patients in Assuit University Trauma Hospital
Brief Title: Sarcopenia and Its Associated Factors Among Hip Fractures Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHAbdelhafeez, resident doctor, Assiut University
Other Study IDs: sarcopenia and hip fracure
Record Dates: First submitted 2021-09-20; First posted 2021-12-02 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Sarcopenia
Keywords: sarcopenia and hip fracture
MeSH Terms: conditions — Sarcopenia; Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: inbody device — measure muscle mass

SUMMARY:
1. Asses the prevalence of sarcopenia in hip fracture patients in Truama hospital at Assuit University
2. To study the associated factors of sarcopenia in hip fracture patients in Trauma hospital at Assuit University

DETAILED DESCRIPTION:
Skeletal muscle is the largest body compartment in most adults with the exception of an enlarged adipose tissue mass in the presence of obesity. Skeletal muscles grow in size from birth onward, reaching peak mass in the third decade. Many factors determine an individual adult's total body skeletal muscle mass and include their size(height),magnitude of adiposity, race, genetic factors, activity, hormone levels and diet. By the fourth decade populations and individuals begin to show a gradual loss in skeletal muscle mass and the rate of atrophy appears to accelerate beyond the seventh decade. The senescence-related changes in skeletal muscle are, in turn, associated with adverse out- comes such as pathological bone fractures and even death. The term sarcopenia, from the Greek roots is widely used to describe the age-associated decrease in muscle mass observed in several cross-sectional and longitudinal studies. Interest in sarcopenia mainly results from its linkage with unfavorable outcomes, including mobility disorders, increased risk of falling, reduced ability to function in activities of daily living, loss of independence, poor quality of life, and reduced life expectancy. Measuring skeletal muscle mass, composition, strength and physical performance is thus a vital part of not only studying sarcopenia, but also of growing importance in clinically evaluating and monitoring the greatly increasing population of ageing at risk adults in most countries. Our report highlights aspects of evaluating these features of skeletal muscle and expands on earlier methodological and historical reviews. While the main phenotypic feature of sarcopenia is loss of lean tissue, notably skeletal muscle, there is growing recognition that sarcopenia can co-exist in the presence of obesity. A skeletal muscle compartment reduced in mass may thus be masked by the presence of excess fat. Diagnosing sarcopenia-obesity may thus include measures beyond that of skeletal muscle mass such as BMI and total body fat, topics that we will allude to in the review that follows. Loss of skeletal muscle also plays an important role in two other conditions, cachexia and frailty, creating a spectrum of phenotypes and clinical conditions that encompass sarcopenia There are two main factors for Skeletal muscle evaluation, skeletal muscle mass and composition, are the main determinants of global muscle metabolic function, strength and physical performance. Vascular and neurological integrity are also essential components that ultimately contribute to a skeletal muscle's metabolic and mechanical functionality. The'quality' of a skeletal muscle is a loosely defined concept that broadly includes aspects of anatomic structure, chemical composition and metabolic and mechanical performance. Our review encompasses aspects of measuring skeletal muscle mass, composition and function in relation to the evaluation of individuals and groups for the presence of sarcopenia and related conditions. Multiple methods of measuring skeletal muscle mass are available for research and clinical purposes that vary in cost, complexity and availability. A high prevalence of low muscle mass in hip-fracture patients has been shown. Hip fractures carry a high risk of both death and disability with a 8-36 % excess mortality within 1 year and more than 50 % of the survivors not regaining their own pre-injury level of independence. Sarcopenia may worsen the functional prognosis after hip fracture occurrence, but the association between reduced muscle mass and functional ability remains unclear in this group of older and frail persons. Conversely, muscle strength has been indicated as a strong independent predictor of the functional outcome, whereas lower-limb performance is usually not accessible at an early stage, because of the direct consequences of the hip fracture on ambulation. There are no available studies in our locality about sarcopenia and its related factors

ELIGIBILITY:
Inclusion Criteria:

* old patients >50 years with hip fracture attending assuit university hospital

Exclusion Criteria:

1. patients with dementia ,muscle disease and neurological disease
2. Patients who are unwilling to participate
3. Patients>80 years due to uncooperate at this age to answer the questionnaire

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: admitted patients in Assiut university Trauma hospital
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sarcopenia among Hip fracture patients in Assuit University Truama hospital | 20 minutes
  by inbody device

CONTACTS AND LOCATIONS:
Overall Officials: Osama Ahmad, prof, Study Chair — assuit yniversity
Locations (1):
- Assiut University, Asyut, Egypt